CLINICAL TRIAL: NCT05013944
Title: AnovaOS Network Powered Patient Registry
Status: Recruiting | Type: Observational
Sponsor: Anova Enterprises, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ANOVA-001-NPPR
Record Dates: First submitted 2021-08-18; First posted 2021-08-20 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Infectious Disease; Neoplasms; Diseases of the Blood and Blood-Forming Organs and Certain Disorders Involving the Immune Mechanism (D50-D89); Endocrine, Nutritional and Metabolic Diseases (E00-E89); Mental and Behavioural Disorders; Diseases of the Nervous System; Diseases of the Eye and Adnexa; Diseases of the Ear and Mastoid Process; Diseases of the Circulatory System; Diseases of the Respiratory System; Diseases of the Digestive System; Diseases of the Skin and Subcutaneous Tissue; Diseases of the Musculoskeletal System and Connective Tissue; Diseases of the Genitourinary System; Pregnancy, Childbirth and the Puerperium; Certain Conditions Originating in the Perinatal Period; Congenital Malformations, Deformations and Chromosomal Abnormalities (Q00-Q99); Symptoms, Signs and Abnormal Clinical and Laboratory Findings, Not Elsewhere Classified; Injury, Poisoning and Certain Other Consequences of External Causes; External Causes of Morbidity and Mortality; Factors Influencing Health Status and Contact With Health Services
Keywords: infectious disease, cancer/oncology, neurology, immunology, cardiology
MeSH Terms: conditions — Communicable Diseases; Neoplasms; Metabolic Diseases; Mental Disorders; Nervous System Diseases; Eye Diseases; Ear Diseases; Respiration Disorders; Digestive System Diseases; Skin Diseases; Urogenital Diseases; Congenital Abnormalities; Chromosome Aberrations; Wounds and Injuries; Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is the development, implementation and management of a registry of patient data that captures clinically meaningful, real-world, data on the diagnosis, nature, course of infection, treatment(s) and outcomes in patients with complex disease globally.

DETAILED DESCRIPTION:
The AnovaOS™ Network Powered Patient Registry may be used to inform the development and conduct of clinical trials and observational studies designed to better understand, prevent, diagnose, treat, ameliorate or cure disease. The AnovaOS™ Network Powered Patient Registry may additionally be used to expedite identification and recruitment of participants for clinical trials of promising therapeutics and observational studies.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older;
* Confirmed positive diagnosis of disease, condition or disorder. This will be self-reported or reported by the patient's provider, advocacy group or other patient representative;
* Laboratory or other independent means of confirmation is not required but may be confirmed in clinical trials;
* Able to understand and willing to sign the informed consent document; or whose legal representative has given consent to participate in the research per state and Federal requirements;
* Willing and able to complete the registry questions or have the instrument(s) completed by an informed proxy;
* Anticipated additional follow up with the registry once per year.

Exclusion Criteria:

* Subjects who do not meet the inclusion criteria for the study;
* Subjects who are unable to understand the protocol or unable to provide legally effective informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Real-world clinical data about patients with complex, serious or immediately life-threatening disease collected as part of the AnovaOS™ platform is important to the scientific community. These data support biopharmaceutical companies, academic researchers and other sponsors with program design and prioritization, study activation and enrolment, and study conduct to help advance promising new therapeutic approaches. Learning from real-world evidence can help inform drug development and help as our research system evolves from a traditional model to one capable of recognizing the benefits of precision medicine.
  The objective of this study is the development, implementation and management of a registry of patient data that captures clinically meaningful, real-world, data on the diagnosis, nature, course of infection, treatment(s) and outcomes in on patients with complex disease globally.
Sampling Method: Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Assess Natural history | 5 years
  Assessing natural history, including estimating the magnitude of a problem; determining the underlying incidence or prevalence rate of a condition; examining trends of disease over time; assessing service delivery and identifying groups at high risk; and describing and estimating survival;
Assess Clinical, Cost and/or Comparative Effectiveness | 5 years
  Determining clinical effectiveness, cost effectiveness, or comparative effectiveness of a test or a treatment;
Assess Safety | 5 years
  Measuring and monitoring safety and harm associated with the use of specific products and treatments, including conducting comparative evaluation of safety and effectiveness;
Measuring and/or Improving Quality of Care | 5 years
  Measuring or improving quality of care, including conducting programs to measure and/or improve the practice of medicine and/or public health.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Walsh, Study Director — Anova Enterprises, Inc; Christopher Beardmore, Principal Investigator — Anova Enterprises, Inc
Locations (1):
- Anova Enterprises, Inc., Arlington Heights, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Further Registry Information — https://anovaevidence.com/
- See also: Registry Sign up — https://anovaevidence.com/